CLINICAL TRIAL: NCT04574323
Title: Short-term Effects of a Paleolithic Lifestyle Intervention in Breast Cancer Patients Undergoing Radiotherapy: A Pilot and Feasibility Study
Brief Title: Effects of a Paleolithic Lifestyle Intervention in Breast Cancer Patients Undergoing Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MVZ Leopoldina GmbH (Other)
Responsible Party: Principal Investigator, Dr. Rainer Klement, Principle investigator, MVZ Leopoldina GmbH
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2020-09-09; First posted 2020-10-05 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Body Weight Changes
Keywords: Bioimpedance analysis; Body composition; Nutrition; Oncology; Paleolithic diet
MeSH Terms: conditions — Breast Neoplasms; Body Weight Changes; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paleolithic lifestyle group (Experimental): The Paleolithic lifestyle (PL) intervention during radiotherapy consists of daily outdoor walks or bike rides of at least 30 min duration, preferably done at noon to maximize vitamin D production, and the adoption of a Paleolithic diet. For the outdoor activity, patients were told to not use sun screen. The Paleolithic diet prescription emphasized the consumption of fatty meats and organ meats from humanely raised animals, wild-caught fish, eggs, nuts and seeds, algae, spices, vegetables and fruits. Excluded were processed foods, grains of all types, legumes, vegetable oils except for native coconut and olive oil and dairy products except for ghee. No dietary supplements were allowed. Patients were supposed to start the PL intervention at least two days prior to the first irradiation and to protocol their food consumption on two days during the first week on the diet. They were also asked about their compliance to the PL intervention at each weekly measurement appointment.
  Interventions: Radiation: Curative radiotherapy; Other: Paleolithic lifestyle intervention
- Standard diet group (Other): This group is on a standard diet while receiving radiotherapy.
  Interventions: Radiation: Curative radiotherapy

INTERVENTIONS:
Radiation: Curative radiotherapy — Standard curative radiotherapy
Other: Paleolithic lifestyle intervention — This intervention consists of daily outdoor walks or bike rides of at least 30 min duration, preferably done at noon to maximize vitamin D production, and the adoption of a Paleolithic diet. For the outdoor activity, patients were told to not use sun screen. The Paleolithic diet prescription emphasized the consumption of fatty meats and organ meats from humanely raised animals, wild-caught fish, eggs, nuts and seeds, algae, spices, vegetables and fruits. Excluded were processed foods, grains of all types, legumes, vegetable oils except for native coconut and olive oil and dairy products except for ghee. No dietary supplements were allowed.
  Arms: Paleolithic lifestyle group

SUMMARY:
The study aims to test the feasibility and effects of a dietary and physical activity intervention based on evolutionary considerations in an oncological setting.

DETAILED DESCRIPTION:
A total of 13 breast cancer patients referred to our clinic for curative radiotherapy were recruited for this pilot study. The women were supposed to undertake a "Paleolithic lifestyle" (PL) intervention consisting of a Paleolithic diet and daily outdoor activity of at least 30 min duration while undergoing radiotherapy. Body composition was measured weekly by bioimpedance analysis. Blood parameters were assessed before, during, and at the end of radiotherapy. A control group on an unspecified standard diet (SD) was assigned by propensity score matching.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >18 kg/m^2
* Karnofsky performance index >60

Exclusion Criteria:

* Metallic body parts
* Unable to comprehend the intervention

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Dropout rate in the Paleolithic lifestyle intervention group | through study completion, an average of 5 weeks
  Used to measure feasibility. The intervention is rated as feasible if dropout rate is <30%
Longitudinal body composition changes | through study completion, an average of 5 weeks
  Measured on a bioimpedance scale (seca mBCA, seca Deutschland, Hamburg, Germany)
Change in vitamin D levels | through study completion, an average of 5 weeks
  Difference between final (average 5 weekks) and baseline 25-hydroxyvitamin D level

SECONDARY OUTCOMES:
Change in beta-hydroxybutyrate levels | through study completion, an average of 5 weeks
  Change between baseline and final (average 5 weeks) beta-hydroxybutyrate levels

CONTACTS AND LOCATIONS:
Locations (1):
- Leopoldina Hospital Schweinfurt, Department of Radiotherapy and Radiation Oncology, Schweinfurt, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Will be made available upon reasonable request. Plan is also to publish all data of this and the KETOCOMP study (NCT02516501) together as soon as all analyses have been published.
Time Frame: The data can be requested from now on.
Access Criteria: A reasonable request to the study P.I. (Dr. Klement) suffices.

REFERENCES:
- [Result] Klement RJ, Koebrunner PS, Krage K, Weigel MM, Sweeney RA. Short-term effects of a Paleolithic lifestyle intervention in breast cancer patients undergoing radiotherapy: a pilot and feasibility study. Med Oncol. 2020 Nov 28;38(1):1. doi: 10.1007/s12032-020-01443-0. PMID 33247817